CLINICAL TRIAL: NCT04842227
Title: Regional Anesthesia for Cardiac Implantable Electronic Device Implantation
Brief Title: Blocks Alternative to Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Habib Khan (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Sponsor-Investigator, Habib Khan, Assistant Professor in Cardiology, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10942
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Pacemaker Implantation; ICD Implantation
MeSH Terms: interventions — Nerve Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Nerve block — Step 1: A small amount of local anesthetic (3-5cc of 0.5% ropivacaine) is administered under ultrasound guidance in the area of the supraclavicular nerve at the base of the neck under sterile conditions. This provides dense anesthesia of the skin and eliminates the need to introduce larger quantities of local anesthetic directly to the skin around the incision (usually 20mL).
  The second step involves introducing 10-15cc of 0.5% ropivacaine under ultrasound guidance into the compartment between the pectoralis major and minor muscles to anesthetize the medial and lateral pectoral nerves. NOTE: Usual care involves "blind" administration of local anesthetic diffusely to the tissues in this region without targeting any particular nerves, and requires larger volumes of anesthetic (40mL for the "blind approach" vs 10-15mL for the nerve block).

SUMMARY:
Current practice is to implant cardiac electronic devices using intravenous sedation with midazolam and fentanyl, as well as local injection of anesthetic (1-2). However, some patients do not tolerate sedation and develop nausea/vomiting, delirium/confusion, allergic reactions, and hemodynamic instability with sedation (2-4). Many patients are poor candidates for procedural sedation due to inadequate fasting before the procedure or prior adverse effects of procedural sedation. Pain control is usually adequate, but a large portion of patients still experience pain or discomfort at the implant site if the local anesthetic did not reach every component of the tissue in the surgical field. Meanwhile, nerve block procedures have been used for decades to improve peri-operative and post-operative pain and reduce sedation requirements. With the introduction of ultrasound, the investigators are able to direct delivery of local anesthetic to anesthetize the supraclavicular and pectoralis nerves that supply sensory/pain sensation to the surgical site. Similar techniques have been well described as safe and effective (5-10). The investigators hypothesize this will improve pain control during and after surgery, reduce or eliminate the need for intravenous sedation and improve the safety of the procedure.

DETAILED DESCRIPTION:
Inpatients who are consented to have cardiac device implantation will be given study information as soon as the decision to implant a device is reached. The patients will have time to decide to participate in the study up until they are called for the procedure (2-72 hours, most commonly > 24 hours). The decision to participate in the study is conveyed to the investigator in the holding room, and written consent is obtained if the patient agrees to participate in the study.

The nerve block is performed in the holding room as a 2-step procedure by trained physicians.

After the nerve block approximately 30-60 minutes will be allowed for the anesthetic to take effect prior to the cardiac device implantation procedure. The patient will be monitored by the nurses in the holding room. Once the patient is taken to the operating room and prepped for the cardiac device implantation procedure, testing of the nerve blocks is performed. The superficial pin-prick test will be performed to determine the success of the SCN block, and a deeper test will be performed with a 22ga needle to ensure the deeper muscular layers are anesthetized and the PECs I block is successful. If both blocks are successful, the patient will receive optional light sedation with midazolam 0.01 mg/kg based on their preference, and the procedure can commence. If either the SCN or PECs blocks are not successful based on the sensation test, usual care is provided.

Immediately after the procedure, the patient is asked to rate the pain during the procedure on a numerical scale. Any adverse effects reported by the patient will be documented. The patient will then be reassessed 1 hour after the procedure in the holding room and then called the following day. One of the investigators will contact the patient by telephone on the following day (24hr later), and perform a similar assessment. The assessment will involve inquiring how the patient is feeling, documenting any unintended adverse effects, and asking the patient to rate their pain on a numerical scale.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years old,
2. Undergoing cardiac device implantation in the suprapectoral area of the chest.

Exclusion Criteria:

1. Prior neck surgery ipsilateral to the device implantation site
2. Infection over the injection site
3. BMI ≥ 35
4. Uncooperative patient
5. Patient unable to provide consent
6. Patient has a pre-existing implanted cardiac device in the left chest wall area
7. Device implantation is booked in less than 2 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Acute anesthesia of skin and tissue | 30 minutes after nerve block
  Needle prick test will be used over the subjected area to assess the nerve block. This will be measured as binary outcome (1-yes blocked ; 0 - not blocked). The region of anesthesia will also be measured by using an illustration to demarcate the region of block on the skin. The dermatomal distribution of the block will be measured in cm2.

SECONDARY OUTCOMES:
Pain score | 0 hour of completion of device implant, 1 hour post procedure and 1 day post procedure.
  Pain score analog will be used to quantify the amount of pain during the procedure. Pain analog score is between 1-10 (1 being no pain to 10 being severe pain).
IV sedation and pain | 0 hour
  Quantify amounts(milligram) of additional sedation or pain relief required intravenously during the procedure
Duration of procedure | 0 hour
  Quantify time required to complete the block
Safety of the nerve block | Day 1
  Any associated complications from the nerve blocks will be listed in a enumerated way and added together.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre Res. Inc. (Ont.), London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No